CLINICAL TRIAL: NCT00843661
Title: Coadministration of Ezetimibe With Fenofibrate Versus Pravastatin Monotherapy for the Treatment of Hyperlipidaemia in HIV-infected Patients Receiving Protease Inhibitors: a Randomized, Prospective, Controlled Pilot Study.
Brief Title: Coadministration of Ezetimibe With Fenofibrate Versus Pravastatin Monotherapy for the Treatment of Hyperlipidaemia in HIV-infected Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ospedale di Circolo - Fondazione Macchi (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Anna Maria Grandi, Ospedale di Circolo Fondazione MAcchi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFP01
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Last update posted 2011-08-02 (Estimated); Status verified 2011-07

CONDITIONS: HIV; Hyperlipidemia; HIV Infections
Keywords: Treatment Experienced
MeSH Terms: conditions — Hyperlipidemias; HIV Infections | interventions — Ezetimibe; Fenofibrate; Pravastatin

ARMS (2):
- Ezetimibe and fenofibrate (Experimental)
  Interventions: Drug: ezetimibe; Drug: fenofibrate
- Pravastatin (Active Comparator)
  Interventions: Drug: pravastatin

INTERVENTIONS:
Drug: ezetimibe — 10 mg ezetimibe/day
  Arms: Ezetimibe and fenofibrate
Drug: fenofibrate — 200 mg fenofibrate/day
  Arms: Ezetimibe and fenofibrate
Drug: pravastatin — 40 mg pravastatin/day
  Arms: Pravastatin

SUMMARY:
* The aim of the study is to compare the effects of coadministration of ezetimibe 10 mg/die + fenofibrate 200 mg/die versus pravastatin 40 mg/die monotherapy in HIV-infected patients treated with protease inhibitors.
* Single-centre, open, randomized, controlled, prospective pilot study.
* 60 patients will be enrolled in order to reach the target of 50 patients evaluable at the end of the study. The patients will be randomly assigned to a 6-month treatment with ezetimibe+fenofibrate or with pravastatin.The visit will be every month.

ELIGIBILITY:
Inclusion Criteria:

* patients older than 18 years
* documented positive HIV antibodies test
* on stable therapy with PIs for at least 12 months
* LDL-cholesterol >130 mg/dl or triglycerides 200 - 500 mg/dl with non-HDL cholesterol >160 mg/dl
* unresponsive to dietary measures and regular physical exercise of at

Exclusion Criteria:

* history of dyslipidemia before antiretroviral therapy
* cardiovascular and cerebrovascular diseases
* Cushing's syndrome
* concurrent therapy with lipid-lowering agents, oral anticoagulant, estrogens, thiazidic diuretics, beta-blockers
* hypothyroidism
* Type 1 diabetes mellitus
* renal failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-03; Primary Completion 2011-12 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
per cent changes of LDL cholesterol, comparison between the 2 treatment regimens | After 6 month treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale di Circolo and Fondazione Macchi, Varese, Varese, Italy